CLINICAL TRIAL: NCT04436133
Title: A Randomized, Blind, and Positive Control Design to Evaluate the Immunization Efficacy of 11 Valent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha) in Chinese Women Aged 18-26 Years
Brief Title: Immunogenicity AND Safety Study of the 11 Valent Recombinant Human Papillomavirus Vaccine (Hansenulapolymorpha)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: Chengdu Institute of Biological Products Co.,Ltd. (Industry); Simoon Record Pharma Information Consulting Co., Ltd. (Industry); Guangxi Center for Disease Control and Prevention (Other Government); Beijing Kantorico Statistical Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GXIRB2020-0036
Record Dates: First submitted 2020-06-11; First posted 2020-06-17 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: HPV Infection; HPV-Related Cervical Carcinoma
MeSH Terms: conditions — Papillomavirus Infections | interventions — Biological Products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vaccine group (Experimental)
  Interventions: Biological: Biological/Vaccine: 11-valent recombinant human papilloma virus vaccine (Hansenula polymorpha)
- Positive control group (Active Comparator)
  Interventions: Biological: 9-valent HPV vaccine（Gardasil 9）

INTERVENTIONS:
Biological: Biological/Vaccine: 11-valent recombinant human papilloma virus vaccine (Hansenula polymorpha) — Inject vaccine produced by ChinaVaccineSerum, containing HPV antigen protein, 270μg/1ml per bottle
  Arms: vaccine group
Biological: 9-valent HPV vaccine（Gardasil 9） — Inject Gardasil 9 , containing HPV antigen protein, 270μg/0.5ml per bottle
  Arms: Positive control group

SUMMARY:
A total of 480 Chinese women aged 18-26 years old were enrolle，experimental group and the control group were randomly assigned in a ratio of 3:1. 360 Chinese women in the experimental group and 120 in the control group. All subjects enrolled in the upper arm deltoid muscle were injected with 3 doses of test vaccine or control vaccine according to the 0, 2, and 6 months immunization program.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women aged 18-26 who can provide legal identification;
2. The subject has the ability to understand the research procedure and sign an informed consent;
3. Subjects have the ability to read, understand, fill out diary cards/contact cards and other research application forms and promise to participate in regular follow-up as required by the research;
4. No previous history of HPV vaccination, no participation in HPV vaccine clinical trials, and no plans to receive HPV vaccine during the study period; The subject was not breastfeeding or pregnant (negative urine pregnancy test), did not have a birth plan within 7 months of enrollment; and from day 1 of the last menstrual cycle to day 0 of the study, did not have sex with men or with men Effective contraception was used during sex and no contraceptive failures occurred (examples of contraceptive failure include male condom rupture during sex). And agreed to continue to take effective contraceptive measures within the first 7 months after participating in the study (effective contraceptive measures include: oral contraceptives, hormone patches, intrauterine devices, condoms, cervical caps, etc.).

First dose exclusion criteria:

1. Previous history of cervical lesions (such as abnormal cervical cancer screening, history of CIN disease) or history of hysterectomy surgery (vaginal or total hysterectomy) or history of pelvic radiation therapy; previous history of external genital diseases (such as vulvar epithelium) Neoplasia, intraepithelial neoplasia and genital warts, etc.);
2. Previous history of severe allergic reactions requiring medical intervention for any vaccine or drug (including yeast) (eg: anaphylactic shock, allergic throat edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction) Wait);
3. Immune function is impaired or has been diagnosed with congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile Rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases;
4. Long-term treatment with immunosuppressive agents, such as: long-term (more than 2 weeks in a row) treatment with glucocorticoids (eg, prednisone or similar drugs);
5. Receive any immunoglobulin or blood products within 3 months before vaccination, or plan to receive such products before the 7th month of the study;
6. Received inactivated vaccine or recombinant vaccine within 14 days before vaccination, or received any live vaccine within 28 days;
7. Loss of spleen or functional spleen, and removal of spleen or spleen caused by any situation;
8. Has been diagnosed with a disease that may interfere with the progress or completion of the study, such as: suffering from severe cardiovascular disease (pulmonary heart disease, pulmonary edema), severe liver and kidney disease, diabetes with complications, etc.; or has been diagnosed with Infectious diseases, such as: active tuberculosis, hepatitis B, hepatitis C, etc.;
9. A history of convulsions, epilepsy, encephalopathy, mental illness, family history of mental illness, etc.;
10. There are thrombocytopenia or other coagulation disorders that can be contraindications to intramuscular injection; 11.3 days before the vaccination, suffering from acute disease or in the acute onset of chronic disease or using antipyretic, analgesic and anti-allergic drugs (such as: acetaminophen, ibuprofen, aspirin, loratadine, cetaxidine Tirizine, etc.);

12.Body temperature before inoculation≥37.3℃(armpit body temperature); 13. People who have a systolic blood pressure ≥140mmHg and/or a diastolic blood pressure ≥90mmHg before enrollment; 14. Participate or plan to participate in other clinical trials (drugs, vaccines and medical devices) during the study; 15. Plan to move out of the local area before the end of the study or leave the area for a long time during the scheduled study visit;

Exclusion criteria for second and third doses of vaccination:

1. Before vaccination (the day of vaccination), pregnant or urine pregnancy test (HCG) is positive; Note: If the subject chooses to terminate the pregnancy, at least 6 weeks after the end of pregnancy and the urine pregnancy test is negative on the day before the vaccination, or the medical certificate of termination of pregnancy issued after the end of pregnancy indicates that HCG levels have returned to normal levels, you can continue Vaccination; if you choose to continue pregnancy, you will not be vaccinated for subsequent doses.
2. Newly discovered or newly occurred conditions that meet the first dose exclusion criteria (except Articles 1 and 13);
3. Other serious adverse events: The researcher decides whether to terminate the test vaccination according to his treatment needs;
4. The investigator assessed any other reasons why the vaccination for the trial should be terminated.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Anti-HPV neutralizing antibodies GMT | 30 days after full immunization
Anti-HPV neutralizing antibody positive conversion rate（after full immunization 30 days） | 30 days after full immunization
Collect all SAEs | through study completion, an average of 13 months
  Vaccine-related and unrelated
Collect AEs incidence | Within 30 minutes of injection
  Vaccine-related and unrelated
Collect AEs incidence | Within 30 days after inoculation
  All AEs: incidence of AEs related to vaccines and unrelated
  The rate of Solicited for AE
  Non-collective AEs: incidence of AEs related to vaccines and unrelated
  AE level 3 and above: incidence of vaccine-related and unrelated AEs
collect AEs leading subject to withdrawal | through study completion, an average of 13months
  Incidence of vaccine-related and unrelated AEs
collect All pregnancy conditions and pregnancy outcomes | through study completion, an average of 13 months
  collect pregnant woman Anti-HPV neutralizing antibody positive conversion rate and Anti-HPV neutralizing antibodies GMT

CONTACTS AND LOCATIONS:
Locations (1):
- Liucheng Center for Disease Control and Prevention, Liuchow, Guangxi, China

IPD SHARING:
Plan to Share IPD: No